CLINICAL TRIAL: NCT06886815
Title: The Effects of Popliteal Nerve Block on Pain and Nerve-Related Symptoms After Acute Achilles Tendon Rupture Repair Surgery: A Randomized Controlled Trial
Brief Title: Popliteal Nerve Block for Acute Achilles Tendon Rupture Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-0039-B
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Achilles Tendon Rupture
Keywords: Popliteal Nerve Block; Lower Extremity Regional Anesthesia; Achilles Tendon

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, double-blinded, randomized controlled superiority trial with two parallel arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: As noted above, only the individual administering the intervention will be aware of allocation assignment. The participant and outcomes assessors will be blinded to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Popliteal nerve (PN) block group (Experimental): 30 mL of 0.5% ropivacaine with 2.5 µg/ml of epinephrine
  Interventions: Procedure: Popliteal Nerve Block
- Placebo Nerve Block (Sham Comparator): 1 mL of saline
  Interventions: Procedure: Sham Block

INTERVENTIONS:
Procedure: Popliteal Nerve Block — Under ultrasound guidance, a 22G, 80-mm echogenic needle (SonoTAP II, Pajunk Medical Systems, USA) will be inserted using an in-plane lateral-to-medial approach. 30 mL of 0.5% ropivacaine with 2.5 µg/ml of epinephrine will be deposited between tibial and common peroneal nerves within the paraneural sheath. Adequate spread of local anesthetics will be confirmed by visualization of paraneural spread.
  Other Names: Popliteal Sciatic Nerve Block
  Arms: Popliteal nerve (PN) block group
Procedure: Sham Block — Patients in the Control group will receive sham blocks using a 25G needle to inject 1 mL of saline subcutaneously in the same location (popliteus of the surgical knee). Sterilization and ultrasound scanning will match actual PN block. Such a non-invasive placebo allows maintaining patient blinding, while reducing the risks associated with high-volume placebo nerve block injections. The ultrasound screen will be blinded from the patient's vision for all patients in the trial to prevent unblinding by patients with knowledge of the technique.
  Arms: Placebo Nerve Block

SUMMARY:
Achilles tendon rupture is common, yet the value of popliteal nerve block for postoperative pain control during surgical repair remains uncertain. Despite widespread use, evidence supporting its analgesic effectiveness is limited, and both popliteal nerve block and Achilles tendon repair carry risks of nerve injury. This randomized, placebo-controlled trial will evaluate whether adding a popliteal nerve block to standard systemic analgesia improves postoperative pain and reduces opioid use in patients undergoing acute Achilles tendon rupture repair. Secondary outcomes will examine the incidence and impact of nerve complications on recovery, including return to physical activity and functional performance.

DETAILED DESCRIPTION:
This will be a prospective, double-blinded, randomized controlled superiority trial conducted at Women's College Hospital (WCH). The study aims to enroll 80 patients (40 per group) undergoing ambulatory surgical repair of acute Achilles tendon ruptures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* ASA classification: I - III
* BMI < 35 kg/m2
* Undergoing acute Achilles tendon rupture repair surgery as a day surgery procedure

Exclusion Criteria:

* Pre-existing neurological deficits or peripheral neuropathy in the distribution of the tibial or common peroneal nerves
* Local infection
* Contraindication to regional anesthesia (e.g., bleeding diathesis, coagulopathy)
* History of use of over 30 mg oxycodone or equivalent per day
* Contraindication to any component of a standard multi-modal analgesia
* Allergy to local anesthetics
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Inability to provide informed consent
* Patient refusal of popliteal nerve blockade
* Prior Achilles tendon surgeries on the operative leg
* Unable to speak or read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption | The first 24 hours after surgery
  Total opioid dose administered to each patient, converted to oral morphine equivalents.

SECONDARY OUTCOMES:
Area Under the Curve for Postoperative Pain | The first 24 hours after surgery
  Area under the curve calculated from discrete Numeric Rating Scale evaluations of postoperative pain (0 - 10), where 0 corresponds to no pain, and 10 corresponds to the worst pain imaginable. Pain will be measured on this scale at 0, 6, 12, 18, and 24 hours after surgery.
Quality of Recovery | At baseline, 6, 24, 48 hours, 7 days and 1-year post-surgery
  Quality of recovery evaluated using the QoR-15 scale (0 - 150), where 0 represents extremely poor recovery and 150 represents excellent recovery.
Postoperative Pain Score | At baseline, 0, 6, 12, 18, 24, 36, 48 hours, 7 days and 1-year post-surgery.
  Measured using the Numeric Rating (NRS) Scale (0 - 10) where 0 corresponds to no pain, and 10 corresponds to the worst pain imaginable.
Intraoperative Opioid Consumption | The first 24 hours after surgery
  Measurement of opioids administered during surgery, converted into oral morphine equivalents.
Time to Analgesic Request | The first 24 hours after surgery
  Length of time until the patient's first request for analgesics following surgery.
Time to Discharge | The first 24 hours after surgery
  The length of time each patient stays in Phase I (Postanesthesia Care Unit) and Phase II (Surgical Day Care) after surgery.
Adverse Events Attributable to Popliteal Block | At 0, 6, 12, 18, 24, 36, 48 hours, 7 days and 1-year post-surgery
  The incidence of adverse events possibly attributable to popliteal nerve block, including peripheral nerve injury, hematoma, and infection.
Adverse Events Attributable to Opioids | Evaluated at 24 and 48 hours after surgery.
  The incidence of opioid-related side effects, including sedation, pruritis, nausea/vomiting, and respiratory depression.
Pain, fatigue, and physical function | Prior to surgery and 1-year post-surgery
  Measured using the Achilles tendon Total Rupture Score (ATRS)
Neuropathic pain | At 1 week and 1-year post-surgery
  Measured using the English version of the Douleur Neuropathique 4 (DN4) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brenna CTA, Khan S, Abdallah FW, Brull R. Achilles Hero or Heel? A Systematic Review of Popliteal Nerve Block for Achilles Repair. Foot & Ankle Surgery: Techniques, Reports & Cases. 2025:100474.